CLINICAL TRIAL: NCT03676283
Title: Increasing Preparedness for Caregiving, Death and Continued Life in Partners of Patients With Incurable Cancer - a Webtrial
Brief Title: Increasing Preparedness Through a Website
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ersta Sköndal University College (Other)
Responsible Party: Principal Investigator, Anette Alvariza, Associate professor, Ersta Sköndal University College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ErstaSUC2
Record Dates: First submitted 2018-09-12; First posted 2018-09-18 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Palliative Care
MeSH Terms: interventions — Caregivers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Web-based psycho-educational support for family caregivers (Experimental): Gaining access to the website (närstående.se) with supportive films and texts
  Interventions: Other: Web-based psycho-educational support for family caregivers

INTERVENTIONS:
Other: Web-based psycho-educational support for family caregivers — A website including potentially modifiable topics shown to be associated with preparedness. The topics cover areas such as knowledge about medical issues including symptoms and symptom relief, communication within the couple, how to spend the time before death, being partner or caregiver, planning of the moment of death and considerations of the partner's future, including psychological issues, logistical issues, economy, and the care for children.

SUMMARY:
Partners of patients with advanced cancer often take a great responsibility for the patient's care. They are often unprepared for a situation where they are faced both with the role as caregivers and with the patient's impending death. This project holds significant research questions on how to implement a web-based intervention and make it easily available to all those in need and prevent negative consequences related to caregiving and the loss of a partner. The project will study the effects of using a website for support and information. Instruments for measuring outcomes will be available both on paper or electronically. To obtain data for the main outcomes, preparedness for caregiving and for death, 200 partners will be recruited and receive access to the website. Preparedness for caregiving will be measured at baseline and four weeks later (pre- and post-intervention. Further, sem-structured interviews will be performed. Preparedness for death will be measured eight weeks after the patient's death. Because current trends point towards increased levels of home-care, web-based interventions could be a way to reach more partners in a more cost-effective way.

DETAILED DESCRIPTION:
Partners of patients with advanced cancer often take a great responsibility for the patient's care. They are often unprepared for a situation where they are faced both with the role as caregivers and with the patient's impending death. This lack of preparedness has been associated with psychological and physical unhealth. Interventions delivered by multi-professional palliative care teams have proved to be effective both in promoting preparedness for caregiving, death and the continued life of the bereaved. This project holds significant research questions on how to implement an intervention and make it easily available to all those in need and prevent negative consequences related to caregiving and the loss of a partner. To reach as many partners as possible, a web-based intervention has been developed on a website (närstående.se) which consists of supportive films and text as well as an online forum. The films show conversations between partners (actors) and healthcare professionals (authentic). The conversations concern potentially modifiable topics, such as medical issues and communication, that are associated with preparedness. The project will study the effects of proactive telephone calls that will be delivered to partners with the aim to support their use of the website. Instruments for measuring outcomes will be available both on paper or electronically. To obtain data for the main outcomes, preparedness for caregiving and for death, 200 partners will be recruited and get access to the website. They will also receive a telephone call with instructions on how to use the website and have access to technical support if necessary. Preparedness for caregiving will be measured at baseline and four weeks later (pre- and post-intervention). Preparedness for death will be measured eight weeks after the patient's death. The status of the modifiable topics will be measured at baseline and four weeks later. Physical and psychological health of the partner will be measured one year later. Further, semi-structured interviews will be performed with participants to explore the feasibility and acceptibility of the web intervention. The project will add significant knowledge about whether web-based support has the potential to increase preparedness and decrease negative consequences for partners of patients with advanced cancer during ongoing care and after the patient's death. Because current trends point towards increased levels of home-care, web-based interventions could be a way to reach more partners in a more cost-effective way. This project is meant to be a pilot to a larger study with a randomised controlled design.

ELIGIBILITY:
Inclusion Criteria:

* Being a partner of a patient with a cancer diagnose and a life expectancy of less than 12 months

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Preparedness for caregiving scale | 4 weeks
  Measures family caregivers' readiness to provide care in real time. It consists of eight items measured on a five point scale ranging from 0-5 where higher values indicate better preparedness. The total score ranges from 0-32. No subscales have been reported for this instrument.

CONTACTS AND LOCATIONS:
Overall Officials: Anette Alvariza, PhD, Principal Investigator — Ersta Sköndal Bräcke University College
Locations (1):
- Ersta Sköndal Bräcke University College, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Doveson S, Tibell LH, Arestedt K, Holm M, Kreicbergs U, Alvariza A, Wallin V. Communication about incurable illness and remaining life between spouses and patients with incurable illness receiving specialized home care: effects of a family caregiver-targeted web-based psycho-educational intervention. BMC Palliat Care. 2024 Dec 16;23(1):282. doi: 10.1186/s12904-024-01614-0. PMID 39681862
- [Derived] Alvariza A, Hager-Tibell L, Holm M, Steineck G, Kreicbergs U. Increasing preparedness for caregiving and death in family caregivers of patients with severe illness who are cared for at home - study protocol for a web-based intervention. BMC Palliat Care. 2020 Mar 17;19(1):33. doi: 10.1186/s12904-020-0530-6. PMID 32183803